CLINICAL TRIAL: NCT04821778
Title: Cohort Study of Definitive Chemoradiotherapy for Esophageal or Esophagogastric Junction Cancer
Brief Title: Chemoradiotherapy in Esophageal or Esophagogastric Junction Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2722
Record Dates: First submitted 2021-03-15; First posted 2021-03-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Esophagus Cancer; Esophagogastric Junction Cancer; Chemoradiation; Targeted Therapy; Immunotherapy; Chemotherapy Effect
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Platinum Compounds; Immunotherapy; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Definitive Chemoradiation (Placebo Comparator): This arm received chemoradiation without immunotherapy/targeting agents as definitive treatment.
  Interventions: Radiation: Radiotherapy; Drug: Platinum based chemotherapy; Drug: Paclitaxel based chemotherapy; Drug: 5-FU Analog based chemotherapy
- Chemoradiation Combined With Immunotherapy/targeting agents (Experimental): This arm received chemoradiation with immunotherapy/targeting agents as definitive treatment.
  Interventions: Radiation: Radiotherapy; Drug: Platinum based chemotherapy; Drug: Paclitaxel based chemotherapy; Drug: Immunotherapy; Drug: 5-FU Analog based chemotherapy; Drug: Nimotuzumab

INTERVENTIONS:
Radiation: Radiotherapy — 50-66Gy/1.8-2.2Gy/25-30f
Drug: Platinum based chemotherapy — q1-3W according to physician's preference
Drug: Paclitaxel based chemotherapy — q1-3W according to physician's preference
Drug: Immunotherapy — Anti-PD-1/PD-L1 Antibody
  Arms: Chemoradiation Combined With Immunotherapy/targeting agents
Drug: 5-FU Analog based chemotherapy — W1-5 qW or d1-14, q3W according to physician's preference
Drug: Nimotuzumab — 200-400mg, d1,qW
  Arms: Chemoradiation Combined With Immunotherapy/targeting agents

SUMMARY:
Definitive chemoradiotherapy is the standard of care in unresectable esophageal or esophagogastric cancer. A multidisciplinary approach, including chemotherapy and radiotherapy, is important for these patients. Morerover, molecular targeting agents does not show clear efficacy in EC up to now. Nowadays, the pace of development of cancer immunotherapies is accelerating. Clinical evidence of the efficacy of immune checkpoint inhibitors and adoptive immunotherapies herald the onset of a new era in cancer immunotherapy. There have also been recent developments to provide a promising frontier in extending the use of immunotherpay or targeting agents to radiotherapy. The purpose of this study was to explore the optimal treatment modalities including PD-1/PD-L1 antibody or targeted drug for patients with unresectable esophageal or esophagogastric junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years；
* Esophageal or Esophagogastric cancer；
* Histologically proven squamous cell carcinoma or adenocarcinoma in patients staged as I-IVa(AJCC 8th)；
* Primary treatment performed in Cancer Hospital, Chinese Academy of Medical Sciences；
* ECOG PS score: 0~1；
* Estimated survival time ≥3 months；
* Normal organ and marrow function as defined below:Hemoglobin: greater than or equal to 100g/L ;Leukocytes: greater than or equal to 4,000 G/L; Neutrophil: greater than or equal to 2,000 G/L; Platelets: greater than or equal to 100,000/mm3 ; Creatinine: less than or equal to 1.5 times the upper limit or CCR greater than or equal to 60 ml/min; AST/ALT: less than or equal to 2.5 times the upper limit; Total bilirubin: less than or equal to 1.5 times the upper limit; INR: less than or equal to 1.5 times the upper limit; APTT: less than or equal to 1.5 times the upper limit; PT: less than or equal to 1.5 times the upper limit；
* Informed consent；

Exclusion Criteria:

* With any distant metastasis out of regional lymphatic drainage or in liver, lung, bone, CNS, etc；
* Patients with other cancer history in 5 years except cervical carcinoma in situ and non-malignant melanoma skin cancer；
* Existing active infection such as active tuberculosis and hepatitis；
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia；
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness History of allergic reactions attributed to paclitaxel, albumin or cisplatin；
* Participation in other clinical trials currently or within 4 weeks of selection；
* Pregnant or lactating females；
* Absence of medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2002-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1year
Overall survival | 2 year
Overall survival | 3 year
Overall survival | 5 year

SECONDARY OUTCOMES:
Progression free survival | 1 year, 2 year, 3 year, 5 year
Number of participants with Acute and late toxicities of radiotherapy,chemotherapy and immunotherapy | 3 months
Pathological response rate | 3 months
  Pathological response were classified into three grades.Grade I signifies that there is little shrinkage in the tumor; only mild regression in the tumor cells is observed under themicroscope. Grade II shows gross reduction in size of the tumor and marked regression in the cancer cells microscopically, yet viable nests of cancer tissue are still visible. Grade III implies complete or almost total resolution of the tumor on exploration, and disappearance of the tumor tissue microscopically; only remnants of degenerated cancer cells can be seen (so-called ghost cancer cells).
R0 resection rate | 3 months
Locoregional recurrence free survival | 1 year, 2 year, 3 year, 5 year
Distant metastasis free survival | 1 year, 2 year, 3 year, 5 year

OTHER OUTCOMES:
Analysis of correlation between radiomics signature extracted by LASSO and the number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1 year, 2 year, 3 year, 5 year
Radiomics analysis | 1 year, 2 year, 3 year, 5 year
  Analysis of correlation between radiomics signature extracted by LASSO and the rate of participants who achieve pathological complete response (pCR) and the overall survival based on MRI and CT simulation.
Target dealineation of organs at risk and their impact on the prognosis and adverse effects of radiotherapy | 1 year, 2 year, 3 year, 5 year
Target dealineation of clinical target volumn and their impact on the prognosis | 1 year, 2 year, 3 year, 5 year

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Department 4th of Radiation Oncology, Anyang Cancer Hospital, Anyang, Henan
  - Hunan Cancer Hospital, the Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - Department of Radiation oncology, Jiangsu Cancer Hospital/Jiangsu Institute of Cancer Research/The affiliated Cancer Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Department of Radiation oncology, Jiangsu Province Hospital/The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing

REFERENCES:
- [Derived] Yang X, Wang X, Xiao Q, Ge X, Yu N, Li J, Feng G, Zheng Z, Jiang Y, Lu L, Xia X, Deng L, Zhang T, Wang W, Liu W, Wang J, Xiao Z, Zhou Z, Bi N, Wang H, Chen C, Wang X. Definitive chemoradiotherapy combined with anti-PD-1 immunotherapy for inoperable esophageal squamous cell carcinoma: a multicenter real-world study. Cancer Biol Ther. 2025 Dec;26(1):2504726. doi: 10.1080/15384047.2025.2504726. Epub 2025 May 14. PMID 40367097